CLINICAL TRIAL: NCT03737526
Title: Impact of Anaesthesia Mode on Evaluation of LEEP Specimen Dimensions
Acronym: LEEP-DIM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0050
Record Dates: First submitted 2018-09-17; First posted 2018-11-09 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia
Keywords: loop electrosurgical excision procedure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the influence of anaesthesia (local by cervical block vs. general or spinal anaesthesia) on height and volume of resection specimens in case of conization treatment for cervical intraepithelial neoplasia (CIN).

Prospective observational study of all patients who underwent a first treatment by loop electrosurgical excision procedure (LEEP) for CIN. Height of fresh resection specimens was first measured by the operator and then by the pathologist after formaldehyde fixation. Volume of fresh specimens was measured in a measuring cylinder by fluid displacement.

DETAILED DESCRIPTION:
Measure of conization specimens can be done in the operating theatre on fresh specimen or by pathologist after fixation. Methods and conditions of specimen measurement are rarely, if ever, described in published studies.

To study the influence of anaesthesia (local by cervical block vs. general or spinal anaesthesia) on height and volume of resection specimens in case of conization treatment for cervical intraepithelial neoplasia (CIN).

Prospective observational study of all patients who underwent a first treatment by loop electrosurgical excision procedure (LEEP) for CIN. Height of fresh resection specimens was first measured by the operator and then by the pathologist after formaldehyde fixation. Volume of fresh specimens was measured in a measuring cylinder by fluid displacement.

ELIGIBILITY:
Inclusion Criteria:

* every patient who underwent a first conization procedure
* regardless of indication

Exclusion Criteria:

* patient's refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators conducted a prospective non-randomized controlled study at the Amiens University Hospital (France). The study took place between January and December 2015. The investigators included every patient who underwent a first conization procedure, regardless of indication. The only exclusion criterion was the patient's refusal to participate.Written consent was obtained before procedure. Data was gathered using questionnaires, pre-, per- and post-procedure.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Impact of anaesthesia on height of resection specimens. | 1 year
  evaluate the impact of the excision procedure technique by the mode of anesthesia using the loop electrosurgical on height of resection specimens in case of conization treatment for cervical intraepithelial neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Gondry, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No